CLINICAL TRIAL: NCT06352268
Title: Clinical, Laboratory and Imaging Features, Treatment Trends and Long Term Outcomes of Patients Undergoing Lesioning Procedures for Movement Disorders - A Cohort Study and Registry
Brief Title: Lesioning Procedures for Movement Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Assistant Professor, All India Institute of Medical Sciences
Other Study IDs: IEC-368/17.07.2023
Record Dates: First submitted 2023-09-12; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Dystonia; Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Dystonia; Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lesioning group: Participants who undergo pallidal, subthalamic or thalamic lesioning for the management of Dystonia, Parkinson's disease or essential tremors
  Interventions: Procedure: Pallidal, subthalamic or thalamic lesioning
- Control group: Participants who were considered for pallidal, subthalamic or thalamic lesioning for the management of Dystonia, Parkinson's disease or essential tremors but went on to continue best medical management

INTERVENTIONS:
Procedure: Pallidal, subthalamic or thalamic lesioning — Radiofrequency, ultrasound guided or other lesioning procedures of the Globus pallidus interna, subthalamic nucleus or Vim nucleus of the thalamus for the management of Movement disorders
  Groups: Lesioning group

SUMMARY:
Dystonia is a rare syndrome with varying etiologies. Similarly, tremor conditions refractory to medical management and disabling that they need surgical interventions are rare in our setting. So far there are no randomized controlled trials of pallidotomy for management of dystonia. There is scant literature on the long term efficacy and safety of Pallidotomy, thalamotomy and other such lesioning procedures in the management of movement disorders. The current literature is significantly plagued by publication bias as case reports with successful outcomes are likely to be selectively published in journals or conference abstracts. Lesioning procedures though seem to be effective are often considered to be risky, especially bilateral pallidotomy is not preferred by several centres. However, our center routinely performs simultaneous bilateral pallidotomy. To generate long term data on the efficacy and safety of lesioning procedures in rare diseases like dystonias especially the effect of functional neurosurgery on varying etiologies of the disease, robust registries are required which collect data on all consecutive patients who undergo the procedure.

DETAILED DESCRIPTION:
Introduction Deep brain stimulation surgery (DBS) has become the standard of care for the management of generalized dystonia and Parkinson's disease with motor fluctuations and disabling dyskinesias. It has been shown in Randomized controlled trials to be effective and safe. Since the last 30 years, DBS has been used to treat a variety of patients with dystonias, which are of varying etiologies. It has now become the standard of care for patients with Advanced Parkinson disease with motor fluctuations and dopaminergic drug induced dyskinesias. However, the DBS is an expensive system, needs hardware implantation and regular programming. It is associated with surgical implantation which may lead to complications such as infection of the hardware, leads and electrodes. Since it is expensive, it is out of reach for the majority of the patients who pay out of pocket. It leads to increased healthcare costs because of the initial expenses for the implant as well as regular follow ups for programming. The programming is currently labour intensive and needs long hours of observation with trial and error to find the optimum programming settings for the individual patient. This may need the patient to be admitted in the inpatient setting or multiple outpatient visits for the patient, which can lead to loss of working hours and burden on the healthcare system. Before the introduction of DBS by Benabid, functional neurosurgery with lesioning procedures such as pallidotomy, thalamotomy, subthalamotomy were used to manage movement disorders such as dystonia, tremors and Parkinson disease. However after the advent of DBS, these procedures have taken a backseat. Also there are no randomized trials for the safety and efficacy of lesioning procedures in dystonias. The current practice in various centers of the world is to unilateral pallidotomy in most cases of dystonia. Simultaneous bilateral pallidotomy is not preferred by several practitioners due to the risk of bulbar symptoms which may be irreversible in certain cases. However, our experience in our Institute suggests good outcomes in patients with various forms of focal and generalized dystonias undergoing simultaneous bilateral pallidotomy using radiofrequency ablation. Similarly the investigators have done pallidotomy for genetic dystonias such as NBIAs (Neuronal brain iron deposition), Wilson's disease who had disabling dystonias or medically refractory status dystonicus. However, the long term efficacy and safety of these patients is not clear as there are no registries or long term follow up data. Similarly in Parkinson Disease the investigators have only a handful of patients who underwent Pallidotomy. Systematic data collection in a multicentric registry to generate meaningful information for patients and clinicians help understand the risks and benefits of the procedures and offer relevant information for clinical decision making.

Problem statement Evidence based management requires robust data to make clinical decisions. This data is derived from studies which may be observational or interventional. In the evidence pyramid, meta-analysis of randomized controlled trials is considered to be of the highest quality of evidence. In some conditions due to the high effect size or due to the rarity of the disease, it may be difficult to conduct randomized controlled studies and the current practice is guided by available observational study literature. Dystonia is a rare syndrome with varying etiologies. Similarly, tremor conditions refractory to medical management and disabling that they need surgical interventions are rare in our setting. So far there are no randomized controlled trials of pallidotomy for management of dystonia. There is scant literature on the long term efficacy and safety of Pallidotomy, thalamotomy and other such lesioning procedures in the management of movement disorders. The current literature is significantly plagued by publication bias as case reports with successful outcomes are likely to be selectively published in journals or conference abstracts. Lesioning procedures though seem to be effective are often considered to be risky, especially bilateral pallidotomy is not preferred by several centres. However, our center routinely performs simultaneous bilateral pallidotomy. To generate long term data on the efficacy and safety of lesioning procedures in rare diseases like dystonias especially the effect of functional neurosurgery on varying etiologies of the disease, robust registries are needed which collect data on all consecutive patients who undergo the procedure. The screening log will include all patients who are being considered for lesioning procedures. How long after diagnosis or medical management the patients are referred for surgery is currently unknown. The patients often receive a course of medical management and botulinum toxin injections. However, the duration is variable. Likewise, even after surgical lesioning, the patients are often continued on medical treatment. The additive effects of surgery with supportive care, palliative care referral patterns, usage of other disease modifiying therapy in patients with wilson's disease etc. are currently not known and this cohort study will shed light on these parameters. Similarly it has been found that some of the patients develop recurrence of symptoms following pallidotomy - either due to progression of the disease or due to relapse as the different dystonia networks develop over time. In such cases some patients are evaluated with repeat imaging and may be subjected to second surgery. There is no data regarding re-do surgery, and these treatment trends will be captured in this cohort.

Review of literature Dystonia There are no randomized controlled trials (RCT) to study the efficacy and safety of pallidotomy or thalamotomy in the management of dystonia. The case series and case reports regarding pallidotomy in dystonia describe a heterogenous population of patients who had undergone the procedure. Most of the case series have a bias towards reporting favourable outcomes. The investigators found a meta-analysis of 100 patients who underwent bilateral procedures for dystonia. This meta-analysis described 33 studies with varying indications such as generalized dystonia, dystonic storm and focal dystonias. The majority of the patients had genetic causes of dystonia with DYT1 gene mutation being the most common known genetic cause. Some studies reported a staged bilateral procedures while some simultaneous bilateral pallidotomy. The median time of follow up was 12 months with a range of 2-180 months. This meta-analysis revealed that 8% patients had transient adverse effects while 11% had permanent adverse effects. The commonest adverse effects that were permanent involved bulbar dysfunction with dysarthria anarthria or mutism. Most of the patients had a lasting beneficial effect while 19% patients had relapse of symptoms on prolonged follow up. The time to relapse of symptoms ranged from 3 weeks to 4.5 years. The predictors of response or relapse were not apparent from this meta-analysis. Moreover, why pallidotomy was preferred in contrast to DBS is not clear from the reports. Another case series describing 89 patients who underwent radiofrequency pallidotomy suggested unacceptable rates of complications with bilateral pallidotomy such as medically refractory parkinsonism, dysarthria and dysphagia. However these are retrospective review of data and the adverse effects may have been selectively reported in both unilateral and bilateral cases. In our center 10 children underwent bilateral simultaneous pallidotomy over a 7 year period and it was found that two patients had undergone the procedure for medically refractory status dystonicus and both of them had resolution of the status dystonicus. Two patients with generalized dystonia had recurrence of symptoms over a follow up of 4.5 years while three had a sustained improvement of more than 40% improvement in BFMDRS (Burke Fahn Marsden Dystonia Rating scale).

Parkinson Disease Pallidotomy in Parkinson's disease has been performed since several decades even before the advent of medical management with levodopa was discovered. There are few RCTs which have looked at the effects of pallidotomy in patients with Parkinson Disease. The European academy of Neurology also recommends pallidotomy in the management of Parkinson's disease with motor fluctuations with dyskinesias being the most responsive symptom to therapy. However with the advent of Deep brain stimulation surgery and the widespread adaptation of implantation of the DBS system, lesioning procedures have taken a backseat. The long term effects of pallidal lesioning on motor and non-motor outcomes and the complications have not been systematically studied. Moreover the concerns of psychic akinesia and corticobulbar syndrome with bilateral pallidotomy has discouraged several practitioners from performing the procedure bilaterally. With the advent of non invasive therapies like MR guided focal ultrasound pallidotomy, the interest in radiofrequency pallidotomy is also resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with movement disorders admitted at the Neurology wards/attending clinics
* Who are being considered for lesioning procedures
* Of all ages and sexes

Exclusion Criteria:

· Those who deny consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with movement disorders such as Dystonia, Tremors or Parkinson's Disease who are being considered to undergo pallidal, subthalamic or thalamic lesioning procedures.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Long term functional outcomes | 1 year
  Long term outcomes in patients undergoing lesioning procedures for the treatment of Dystonia - Burke Fahn Marsden Dystonia - Disability scale. Lesser score is better
Long term functional outcomes | 1 year
  Long term outcomes in patients undergoing lesioning procedures for the treatment of Parkinson Disease - Unified Parkinson Disease Rating Scale (UPDRS). Lesser score is better

SECONDARY OUTCOMES:
Predictors of outcomes | 1 year
  To study the factors determining outcomes in patients undergoing lesioning procedures for movement disorders
Demography | Baseline at enrolment
  To study the demographic features (age, gender, age of onset, age at which lesioning is done) of patients undergoing lesioning procedures for the treatment of Movement disorders
Clinical features | Baseline at enrolment
  To study the clinical features in patients undergoing lesioning procedures for the treatment of Movement disorders
Laboratory findings | Baseline at enrolment
  To study the laboratory findings, genetic study results in patients undergoing lesioning procedures for the treatment of Movement disorders
Imaging features | Baseline at enrolment
  To study the imaging features in patients undergoing lesioning procedures for the treatment of Movement disorders
Treatment trends | At baseline
  Treatment trends including medication prescription patterns, pattern of referral to surgery, need for redo surgery
Clinical features | At 1 year
  To study the clinical features in patients undergoing lesioning procedures for the treatment of Movement disorders
Treatment trends | 1 year
  Treatment trends including medication prescription patterns, pattern of referral to surgery, need for redo surgery

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: From end of study to five years later
Access Criteria: To be provided after approaching through Institute Ethics committee, AIIMS New Delhi